CLINICAL TRIAL: NCT01491698
Title: A Pilot Randomized Controlled Trial Examining the Impact of Roux-En-Y Pouch Reconstruction Compared With Conventional Roux-En-Y Reconstruction on Health-Related Quality of Life in Patients Undergoing Total Gastrectomy for Adenocarcinoma
Brief Title: Impact of Roux-En-Y Pouch Reconstruction Compared With Conventional Roux-En-Y Reconstruction on Health-Related Quality of Life in Patients Undergoing Total Gastrectomy for Adenocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-070
Record Dates: First submitted 2011-12-09; First posted 2011-12-14 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Gastric Cancer
Keywords: stomach; surgery; Total Gastrectomy; Roux-En-Y Pouch Reconstruction; Conventional Roux-En-Y Reconstruction; Quality of Life; 11-170
MeSH Terms: conditions — Stomach Neoplasms | interventions — Pliability; Postoperative Period

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- pts undergoing Roux-en-Y pouch reconstruction (RYP) (Experimental): This is a pilot randomized controlled trial comparing changes in health-related quality of life (HRQOL) in patients undergoing Roux-en-Y pouch reconstruction (RYP) with patients undergoing conventional Roux-en-Y reconstruction (RYC) following total gastrectomy for adenocarcinoma.
  Interventions: Procedure: Roux-en-Y pouch reconstruction (RYP)
- pts undergoing conventional Roux-en-Y reconstruction (RYC) (Active Comparator): This is a pilot randomized controlled trial comparing change in health-related quality of life (HRQOL) in patients undergoing Roux-en-Y pouch reconstruction (RYP) with patients undergoing conventional Roux-en-Y reconstruction (RYC) following total gastrectomy for adenocarcinoma.
  Interventions: Procedure: conventional Roux-en-Y reconstruction (RYC)

INTERVENTIONS:
Procedure: Roux-en-Y pouch reconstruction (RYP) — Patients will be consented to the study and complete pre-surgical questionnaires. Final randomization will occur once the surgeon in the operating room has confirmed eligibility intraoperatively. The envelope will be opened, and the patient randomized to either receive RYP or RYC. There are no restrictions on how surgeons may create the RYC or RYP reconstruction, except that the pouch must be a minimum of 15 cm in length (from esophago-jejunal anastomosis to end of jejuno-jejunal anastomosis).
  Other Names: Patients will be seen in follow-up at intervals congruent with routine post-operative; care: post-operative (approximately 1 month), 3 months, 6 months, 12 months,; and 24 months following surgery (+- one month at each time interval to allow; flexibility in scheduling). At each of these visits patients will complete the; HRQOL questionnaires, which require approximately 30 minutes total.
  Arms: pts undergoing Roux-en-Y pouch reconstruction (RYP)
Procedure: conventional Roux-en-Y reconstruction (RYC) — Patients will be consented to the study and complete pre-surgical questionnaires. Final randomization will occur once the surgeon in the operating room has confirmed eligibility intraoperatively. The envelope will be opened, and the patient randomized to either receive RYP or RYC. There are no restrictions on how surgeons may create the RYC or RYP reconstruction, except that the pouch must be a minimum of 15 cm in length (from esophago-jejunal anastomosis to end of jejuno-jejunal anastomosis).
  Other Names: Patients will be seen in follow-up at intervals congruent with routine post-operative care:; post-operative (approximately 1 month), 3 months, 6 months, 12 months, and; 24 months following surgery (+- one month at each time interval to allow flexibility in scheduling). At each of these visits patients will complete the; HRQOL questionnaires, which require approximately 30 minutes total.
  Arms: pts undergoing conventional Roux-en-Y reconstruction (RYC)

SUMMARY:
This study is being done to learn more about how different surgery procedures bring back the eating pathway after removing the stomach in patients with stomach cancer. If the surgeon has decided that some, or all, of the patient's stomach must be removed the surgeon must create a new way to allow food to travel from the mouth to the intestines. Some patients develop problems because they are missing their stomach, such as lack of hunger, bloating, cramping, and heartburn.

The surgeons at Memorial Sloan-Kettering Cancer Center are conducting a study to determine if a change in surgery can help reduce these symptoms.

The most common method of creating a way for food is called a "Roux-en-Y", in which one part of the intestine is connected with the end of the esophagus (the swallowing tube) in the abdomen, and another connection is made between the intestines lower down.

The change in surgery involves creating a pouch from a part of the intestines to replace the stomach.

This study will compare the effects, good and/or bad, of gastric pouch reconstruction with the usual reconstruction to see if the pouch makes you feel better overall.

This type of surgery has been used by some surgeons for many years and is known to be safe, but it is not known if it reduces symptoms or improves nutrition compared with the usual surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Pathologically confirmed gastric adenocarcinoma at MSKCC (biopsy may be performed at other institutions but slides must be confirmed at MSKCC, as is routine care at our institution)
* No evidence of metastases(a)
* Total gastrectomy performed(b)
* Pouch reconstruction is technically feasible(c)

  * Patients will be registered and consent obtained, if the surgeon believes there is no evidence of metastases. If metastatic disease is identified at the time of operation, the patient will not be randomized.
  * Patients will be conditionally enrolled, and consent obtained, if the surgeon believes the patient may need a total gastrectomy at the time of operation. If a total gastrectomy is not performed, the patient will not be randomized.
  * Patients will be excluded if, at the time of surgery, the surgeon feels that creation of a pouch is not technically feasible. This may be due to prior abdominal surgery, anatomic variants, or anything else at the surgeon's discretion.

Exclusion Criteria:

* Not expected to be able to provide follow-up over 2 years (due to geographic or other limitations)
* Not able to complete HRQOL instruments on their own (non-English speaking or physical status)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
feasibility | 2 years
  of recruiting patients with gastric adenocarcinoma to this randomized controlled trial (RCT). We will assess this based on the number of patients who are randomized during the pilot study.

SECONDARY OUTCOMES:
change in HRQOL ( Health-Related Quality of Life) | 2 years
  from preoperative following total gastrectomy, as measured with the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 and QLQ-STO22 questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Coit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/